CLINICAL TRIAL: NCT04640597
Title: A Prospective, Multicentre Observational Study to Evaluate the BioMimics 3D Vascular Stent System in the Treatment of Peripheral Arterial Disease: MIMICS-3D-USA
Brief Title: MIMICS-3D-USA Registry Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Veryan Medical Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: MIMICS-3D-USA
Record Dates: First submitted 2020-11-13; First posted 2020-11-23 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Peripheral Arterial Disease
Keywords: PAD; PVD; SFA stent; stent; Helical stent; Vascular stent
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: BioMimics 3D Vascular Stent System — Patients with BioMimics 3D Vascular Stent System

SUMMARY:
The MIMICS-3D-USA Study is a prospective, multicentre, observational study (non-investigational) of the BioMimics 3D Vascular Stent System that evaluates evaluate safety, effectiveness and device performance within a real-world clinical population of patients undergoing femoropopliteal intervention for the treatment of peripheral artery disease.

DETAILED DESCRIPTION:
The MIMICS-3D-USA Study is designed to enable the collection, analysis, reporting and presentation of data from use of the BioMimics 3D Vascular Stent System purchased by the hospital / institution or office interventional suite and used in accordance with the IFU associated with the product's FDA approval. The intent of this post-market observational study is to increase the understanding of the performance of the BioMimics 3D Vascular Stent System in a larger population of patients representative of a real-world situation within US hospitals, institutions and office-based interventional suites or labs.

ELIGIBILITY:
Inclusion Criteria:

* Patient is age ≥18 and ≤85 years at the date of consent.
* Patient has provided written informed consent for participation in the study prior to index procedure.
* Patient has documented symptomatic peripheral arterial disease scheduled for treatment with the BioMimics 3D Vascular Stent System in accordance with the IFU.

Exclusion Criteria:

* Patients whose lesions cannot be crossed with a wire and/or balloon catheter and cannot be dilated sufficiently to allow passage of the delivery system.
* Patients with a history of intolerance or adverse reaction to antiplatelet and/or anticoagulation therapies, bleeding diathesis or severe hypertension.
* Patients with known hypersensitivity to nickel-titanium.
* Patient has a comorbidity that in the Investigator's opinion would limit life expectancy to less than 12 months.
* Patient is pregnant or breastfeeding.
* Patient is unable or is unwilling to comply with site standard of care procedures

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who receive treatment with Veryan's BioMimics 3D Vascular Stent System in accordance with the current approved FDA (PMA # 180003 approval) indication for use as stated in the Instructions for Use (IFU) will be consecutively enrolled in this study
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2023-09-04 (Estimated); Study Completion 2025-09-04 (Estimated)

PRIMARY OUTCOMES:
Safety endpoint of number of subjects of freedom from CEC-adjudicated major adverse events (MAE) comprising death, any unplanned major amputation performed on the index limb or clinically driven target lesion revascularization (CDTLR) through 30 days. | 30 Days
  Freedom from major adverse events expressed as a percentage
Primary effectiveness endpoint of number of subjects of freedom from CEC Adjudicated clinically driven target lesion revascularization (CDTLR) through 12 months | 12 months
  Freedom from CDTLR at 12 Months expressed as a percentage

SECONDARY OUTCOMES:
Technical success defined as delivery and deployment of the study stent to achieve a final residual diameter stenosis of ≤30% measured by visual assessment of angiographic imaging at the end of the study procedure on Day 0. | Procedural
  Number of participants with final residual stenosis ≤30%
Procedural success defined as technical success with absence of MAE (comprising death, | 24 hours after index procedure
  Number of participants with acute technical success and absence of MAE
Incidence of components of CEC-adjudicated MAE. | 30 days, 12, 24 and 36 months
  Incidence of individual components of CEC-adjudicated MAE (death, any unplanned major amputation performed on the index limb or CDTLR).
Overall rate and incidence of adverse events | 36 Months
  Overall rate and incidence of adverse events from Day 0 to completion of study follow-up at month 36
Primary Stent Patency rate determined by core lab adjudicated, duplex ultrasound at 12 Months | 12 Months
  Primary Stent Patency expressed as a percentage
Comparison of mean Rutherford Clinical Category measured at Baseline, Day 30, Months 12, 24 and 36. | Baseline, Day 30, Months 12, 24 and 36.
  Compare RCC at each of the follow-up visit with the Baseline
Functional outcome: ankle brachial index measurement comparison | Baseline, within 30 days after index procedure, then at Month 12.
  Comparison of the ankle brachial index (ABI) measurement at Baseline, within 30 days after index procedure, then at Month 12.
Comparison of the quality of life (QoL) score at Baseline, within 30 days after index procedure, then at Months 12, 24 and 36 | Baseline, Day 30, Months 12, 24 and 36.
  Compare the change in QoL score compared to the Baseline
Incidence of stent fractures | 36 Months
  Incidence of reported stent fracture reported by investigational sites through 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Nuwani Edirisinghe, Study Director — Veryan Medical
Locations (27):
- United States (27):
  - Alabama Clinical Therapeutics, LLC, Birmingham, Alabama
  - Cardiovascular Associates of the Southeast, Birmingham, Alabama
  - Pulse Cardiovascular Institute, Scottsdale, Arizona
  - Vascular Care Connecticut, Darien, Connecticut
  - Cardiovascular Solutions Institute, Bradenton, Florida
  - Palm Vascular Centers, Miami Beach, Florida
  - Coastal Vascular & Interventional, PLLC, Pensacola, Florida
  - Midwest Cardiovascular Research Foundation, Davenport, Iowa
  - Coastal Vascular & Interventional, PLLC, Davenport, Iowa
  - University of Iowa, Iowa City, Iowa
  - CIS Clinical Research Corporation, Houma, Louisiana
  - Vascular Care Group, Wellesley, Massachusetts
  - University of Missouri, Columbia, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - NJ Endovascular and Amputation Prevention, LLP, Clifton, New Jersey
  - Cardiac And Vascular Interventions of NJ, New Brunswick, New Jersey
  - Columbia University Irving Medical Center/NYPH, New York, New York
  - Columbia University Medical Center, New York, New York
  - Amputation Prevention Center of North Carolina, Cary, North Carolina
  - Advanced Cardiovascular Solutions, Oklahoma City, Oklahoma
  - US cardiovascular of Greenburg, Jefferson Hills, Pennsylvania
  - Ascension Seton Heart Institute, Austin, Texas
  - Cardiothoracic and Vascular Surgeons, Austin, Texas
  - Baylor St Lukes Medical Center, Houston, Texas
  - North Dallas Research Associates, McKinney, Texas
  - Hurricane Cardiology Research, New Braunfels, Texas
  - AZH Wound & Vascular Center, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No